CLINICAL TRIAL: NCT04651257
Title: Role of Contrast Enhanced Digital Mammography in Female Patients With Pathological Nipple Discharge
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Marwa Mohamed Mosaad, principle investigator, Assiut University
Other Study IDs: CEM in nipple discharge
Record Dates: First submitted 2020-09-26; First posted 2020-12-03 (Actual); Last update posted 2020-12-03 (Actual); Status verified 2020-11

CONDITIONS: Contrast Mammography in Pathological Nipple Discharge

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Contrast mammography (CEM) — Contrast mammography in pathological nipple discharge

SUMMARY:
To evaluate the validity of contrast enhanced digital mammography in evaluation of pathological nipple discharge .

DETAILED DESCRIPTION:
Nipple discharge is a relatively frequent complaint in females, being the third most common breast symptoms prompting medical care, after breast pain and breast palpable mass. Over 80% of females will have an episode of nipple discharge during their fertile life,which can be categorized as lactional which is milky in nature and occur during pregnancy or breast feeding. Physiological nipple discharge, is yellow, milky or greenish in nature, it cannot happen spontaneously and it can often be seen coming from multiple orifices,Some causes of physiological nipple discharge are hypothyroidism and medication side-effects. . Pathological nipple discharge is defined as a clear, serous, or bloody secretion , spontaneous, discharging from a single duct and unilateral. It is frequently caused by a benign lesion, such as intraductal papilloma (35-56%) or ductal ectasia (6-59%), but an underlying malignancy can be present in a percentage of cases reported to be variable from 5 to 33%.

Majority of nipple discharge cases are more frequently due to benign conditions, so less operative ,nonsurgical methods can be applied to limit the need for surgical intervention , the woman that presents with nipple discharge should be managed as follow , ultrasound which is always performed in cases with nipple discharge for detection of ductal carcinoma in situ or invasive carcinoma , the sensitivity and specificity of ultrasound were 65% and 75% to 85%respectively ,mammography which plays an important role in diagnosis of breast diseases however it has low (20-25%)sensitivity in cases with nipple discharge as the associated lesions are usually retro areolar ,small, intraductal and non calcified so negative mammography do not exclude the possibility of underlying disease , ductography,which has long been considered the gold standard for evaluation of nipple discharge but it has low sensitivity , MRI has high sensitivity in evaluation of nipple discharge up to 88% to 95%, and its negative predictive value is (90%) , demonstrate not only ductal lesions but also lesions in adjacent parenchyma and it is superior in assessment of location and extent of a lesion.

Recently, contrast enhanced digital mammography has shown a very high sensitivity and specificity in diagnosis of breast lesions, it was approved by the U.S. Food and Drug Administration in 2011. The utility of CEM in the diagnostic setting for evaluation of breast lesion is 100% sensitivity, 87.7% specificity, 76.2%, positive predictive, 100%negative predictive .CEM has been found to result in more accurate tumor size estimation . In the evaluation of suspicious micro calcifications, the negative predictive value of CEM has been reported to be up to 93% . The literature also suggests that the improved performance of CEM relative to that of mammography is greater in women with dense breast tissue as compared with nondense breast tissue, with fewer false-negative cases . Additionally CEM can evaluate response to neoadjuvant chemotherapy and assessment of disease recurrence and also in screening of high risk women .

ELIGIBILITY:
Inclusion Criteria:

1_in diagnosis of female patients with pathological nipple discharge

Exclusion Criteria:

* 1. Patients with renal failure or with raised renal chemistry 2-patients who are allergic to contrast 2. Pregnant women

Ages: 20 Years to 80 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: This study will include 40 patients with pathological nipple discharge
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2020-12 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
To correlate results of CEM with histopathology (TCNB,FNAC,surgical excision) in female patients with pathological nipple discharge . | Baseline
  Pathological nipple discharge has several causes ,inflammatory ,malignant ,benign lesion , this will be evaluated by CEM and correlate the results with histopatholgy of the cases .

REFERENCES:
- [Background] Morrogh M, Park A, Elkin EB, King TA. Lessons learned from 416 cases of nipple discharge of the breast. Am J Surg. 2010 Jul;200(1):73-80. doi: 10.1016/j.amjsurg.2009.06.021. Epub 2010 Jan 15. PMID 20079481
- [Background] Lippa N, Hurtevent-Labrot G, Ferron S, Boisserie-Lacroix M. Nipple discharge: The role of imaging. Diagn Interv Imaging. 2015 Oct;96(10):1017-32. doi: 10.1016/j.diii.2015.07.004. PMID 26433322
- [Background] Ashfaq A, Senior D, Pockaj BA, Wasif N, Pizzitola VJ, Giurescu ME, Gray RJ. Validation study of a modern treatment algorithm for nipple discharge. Am J Surg. 2014 Aug;208(2):222-7. doi: 10.1016/j.amjsurg.2013.12.035. Epub 2014 Apr 3. PMID 24767970
- [Background] Boisserie-Lacroix M, Adenet C, Trillaud H. [Evaluation of suspicious nipple discharge with MRI: review of 50 cases]. J Radiol. 2011 May;92(5):412-20. doi: 10.1016/j.jradio.2011.03.003. Epub 2011 May 7. French. PMID 21621107